CLINICAL TRIAL: NCT00232908
Title: An Open-label Study of a HAART (Highly Active Antiretroviral Therapy) Regimen Containing Subcutaneous Injection of Fuzeon on Quality of Life in Clinically Stable, Treatment-experienced Patients With HIV-1 Infection
Brief Title: QUALITE Study - A Study of Fuzeon (Enfuvirtide) in Treatment-Experienced Patients With Human Immunodeficiency Virus-1 (HIV-1) Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18018
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ARV regimen; Drug: enfuvirtide [Fuzeon]

INTERVENTIONS:
Drug: ARV regimen — As prescribed
Drug: enfuvirtide [Fuzeon] — 90mg sc bid for 12 weeks

SUMMARY:
This study will evaluate patient quality of life and tolerability of a HAART (highly active antiretroviral therapy) regimen containing twice-daily subcutaneous injections of Fuzeon in clinically stable, treatment-experienced patients with HIV-1 infection. All patients will use a 31-gauge thin-walled 8mm needle to administer Fuzeon. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adults or adolescents at least 16 years of age;
* HIV-1 infection;
* clinically stable, treatment-experienced;
* evidence of HIV-1 replication despite ongoing antiretroviral therapy;
* CD4 + count greater than 50 cells/mm3.

Exclusion Criteria:

* previous use of Fuzeon and/or T-1249;
* active, untreated opportunistic infection;
* inability to self-inject, unless a reliable caregiver is available to inject.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2004-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
QoL (MOS-HIV)\n | Baseline and Week 12

SECONDARY OUTCOMES:
Change from baseline in HIV-RNA | Week 12
Change from baseline in CD4 count | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (84):
- United States (81):
  - Phoenix, Arizona
  - Bakersfield, California
  - Berkeley, California
  - Los Angeles, California
  - Modesto, California
  - Oakland, California
  - Palm Springs, California
  - Rancho Mirage, California
  - San Mateo, California
  - Tarzana, California
  - Washington D.C., District of Columbia
  - Bay Pines, Florida
  - Boynton Beach, Florida
  - Brandon, Florida
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - North Palm Beach, Florida
  - Oakland Park, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Pompano Beach, Florida
  - Port Saint Lucie, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - Tallahassee, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Lawrenceville, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Springfield, Illinois
  - Topeka, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Silver Spring, Maryland
  - Berkley, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Butte, Montana
  - Las Vegas, Nevada
  - East Orange, New Jersey
  - Englewood, New Jersey
  - Jersey City, New Jersey
  - Newark, New Jersey
  - Perth Amboy, New Jersey
  - Somers Point, New Jersey
  - West Orange, New Jersey
  - Manhasset, New York
  - Mount Vernon, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Stony Brook, New York
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Portland, Oregon
  - Harrisburg, Pennsylvania
  - Philadelphia, Pennsylvania
  - Reading, Pennsylvania
  - West Reading, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Hampton, Virginia
  - Seattle, Washington
- Puerto Rico (3):
  - Cagaus
  - Ponce
  - San Juan